CLINICAL TRIAL: NCT03223935
Title: A Comparison of Roasted Pulse Snacks on Post-prandial Food Intake, Appetite, and Glycemic Response in Healthy Young Adults
Brief Title: Roasted Pulse Snacks, Post-prandial Food Intake, Appetite, and Glycemia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Collaborators: Saskatchewan Pulse Growers (Other); Pulse Canada (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: HS20792 (B2017:059)
Record Dates: First submitted 2017-07-06; First posted 2017-07-21 (Actual); Last update posted 2023-01-23 (Actual); Status verified 2021-04

CONDITIONS: Normal Weight; Overweight; Normoglycemic
MeSH Terms: conditions — Overweight

STUDY DESIGN:
Intervention Model Description: Randomized, controlled cross-over acute trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Roasted snacks (Active Comparator): Corn nuts
  Interventions: Other: Corn nuts
- Roasted chickpeas (Experimental): Chickpeas
  Interventions: Other: Chickpeas
- Roasted yellow peas (Experimental): Yellow peas
  Interventions: Other: Yellow peas
- Roasted pinto beans (Experimental): Pinto beans
  Interventions: Other: Pinto beans
- Roasted soybeans (Experimental): Soybeans
  Interventions: Other: Soybeans
- Roasted almonds (Experimental): Almonds
  Interventions: Other: Almonds

INTERVENTIONS:
Other: Corn nuts — Roasted corn nut snack
  Arms: Roasted snacks
Other: Chickpeas — Roasted chickpea snack
  Arms: Roasted chickpeas
Other: Yellow peas — Roasted yellow pea snack
  Arms: Roasted yellow peas
Other: Pinto beans — Roasted pinto bean snack
  Arms: Roasted pinto beans
Other: Soybeans — Roasted soybean snack
  Arms: Roasted soybeans
Other: Almonds — Roasted almond snack
  Arms: Roasted almonds

SUMMARY:
An investigation on the effects of roasted pulse snacks on post-prandial glycemic and satiety response in healthy young adults.

DETAILED DESCRIPTION:
An acute, randomized, controlled cross-over trial examining the post-prandial glycemic and satiety response to six snacks will be conducted. The study treatments are: 1) roasted corn nuts, 2) roasted chickpeas, 3) roasted yellow peas, 4) roasted pinto beans 5) roasted soybeans, and 6) roasted almonds. They will be matched for calorie content and provided in 200 kcal servings.

ELIGIBILITY:
Inclusion Criteria:

* BMI: ≥18.5 and ≤29.9 kg/m2
* Fasting serum glucose: ≤5.5 mmol/L

Exclusion Criteria:

* Fasting serum glucose > 5.5 mmol/L
* Smoking
* Thyroid problems
* Previous history of cardiovascular disease, diabetes, liver or kidney disease, inflammatory bowel disease, celiac disease, short bowel syndrome, any malabsorptive syndrome, pancreatitis, gallbladder or biliary disease
* Presence of a gastrointestinal disorder or surgeries within the past year
* Consuming prescription or non-prescription drug, herbal or nutritional supplements known to affect blood glucose or that could affect the outcome of the study as per investigator's judgment
* Known to be pregnant or lactating
* Known intolerance, sensitivity or allergy to any ingredients in the study products.
* Extreme dietary habits (i.e. Atkins diet, very high protein diets, etc.)
* Uncontrolled hypertension (systolic blood pressure ≥140 mm Hg or diastolic blood pressure ≥90 mm Hg)
* Weight gain or loss of at least 10lbs in previous three months
* Excessive alcohol intake
* Restrained Eaters (identified by Eating Habits Questionnaire)

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2017-08-11 (Actual); Primary Completion 2018-04-04 (Actual); Study Completion 2018-04-04 (Actual)

PRIMARY OUTCOMES:
Food intake | At 60 min
  Ab libitum meal

SECONDARY OUTCOMES:
Subjective appetite | 0-200 min
  Measured by VAS questionnaire at 12 time points used to calculate area under the curve
Blood glucose concentrations | 0-200 min
  Measured in blood using a glucometer at 12 time points and used to calculate area under the curve
Physical comfort | 0-200 min
  Measured by VAS questionnaire at 12 time points to calculate area under the curve
Energy and fatigue | 0-200 min
  Measured by VAS questionnaire at 12 time points to calculate area under the curve
Palatability of meal | At 60 min
  Measured by VAS questionnaire
Palatability of treatment | At 5 min
  Measured by VAS questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Peter JH Jones, PhD, Principal Investigator — University of Manitoba
Locations (1):
- Richardson Centre for Functional Foods and Nutraceuticals, University of Manitoba, Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: No
Individual participant data requests should be submitted to the PI.